CLINICAL TRIAL: NCT03043937
Title: Cardiac Diseases With Pregnancy in Benisuef Localities
Status: Completed | Type: Observational
Sponsor: Beni-Suef University (Other)
Responsible Party: Principal Investigator, Momen Zakaria Mohammed mohammed, assisstant lecturer, Beni-Suef University
Other Study IDs: 1200
Record Dates: First submitted 2017-01-06; First posted 2017-02-06 (Estimated); Last update posted 2017-05-19 (Actual); Status verified 2017-05

CONDITIONS: Heart Disease Structural Disorder Abscess of Cardiac Septum
MeSH Terms: interventions — Registries

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- cardiac patients WHO class 1,2
  Interventions: Other: registry
- cardiac patients WHO class 3,4
  Interventions: Other: registry

INTERVENTIONS:
Other: registry

SUMMARY:
The aim of this work is to demonstrate the variation of cardiac diseases among pregnant ladies in our localities, detect maternal & fetal complications and to predict the risk factors for poor maternal, fetal & neonatal outcomes

ELIGIBILITY:
Inclusion criteria

* All pregnant ladies with Cardiac diseases, valvular heart disease, congenital heart disease, ischemic heart disease, cardiomyopathy, arrhythmias , big and pulmonary hypertension, presenting with pregnancy regardless age, any concomitant diseases and type of heart disease will be enrolled.
* A similar number of pregnant females free from previous mentioned cardiac diseases will be studied as controls.

Exclusion Criteria:

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: A prospective analytical study is managed to be commenced in Beni-Suef governorate as cooperation between Department of Cardiology and Department of Obstetrics and Gynaecology Beni-Suef University during the period between Jan/2015 and Dec/2016 among women with cardiac diseases during pregnancy regardless gestational age at presentation and up till 6 weeks postpartum in comparison to women free from any cardiac diseases.
Sampling Method: Non-Probability Sample
Enrollment: 400 (Actual)
Dates: Start 2015-01; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Fetomaternal and neonatal outcome | 2 years
  Number of Participants With abortion,preterm labour,Intrauterine fetal death,Postterm fetus, intrauterine growth restriction,Fetuses with Congenital heart diseases,Neonatal admission to Neonatal Intensive care unit,neonatal death,Perineal,vaginal,broad ligament haematoma, Internal Hemorrhage due to anticoagulant drugs,malfunctioning valve,heart failure ,Thromboembolic complications, perinatal maternal death.

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Medicine, Benisuef, Egypt